CLINICAL TRIAL: NCT01484626
Title: An Open-Label Phase I/II Study of Bendamustine, Weekly Bortezomib, Lenalidomide and Dexamethasone for the Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: Bendamustine, Wkly Bortezomib, Lenalidomide and Dexamethasone for Multiple Myeloma
Acronym: BVRD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Celgene would no longer supply lenalidomide for the study
Sponsor: Loyola University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Scott E Smith, MD, PhD, Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 203145
Record Dates: First submitted 2011-11-28; First posted 2011-12-02 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma; Refractory Multiple Myeloma; Bendamustine; Bortezomib; Lenalidomide; Dexamethasone; Treanda; Velcade; Revlimid
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bendamustine (Experimental): Bendamustine is combined with standard chemotherapy.
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — The first group of three patients to enter the study will receive a 25 mg/m^2 dose of bendamustine. If this dose is found to be safe, the next three patients will receive 50 mg/m^2. Using a modified Fibonacci dose-escalation design, the dose will continue to increase at a rate of 25 mg/m^2 until the highest safe dose of bendamustine is found. The maximum dose will be 125 mg/m^2. Bendamustine and bortezomib will be given through a catheter twice a week every 21 days. Dexamethasone and lenalidomide will be given orally. In general, a cycle of chemotherapy will last 21 days.
  Other Names: Treanda

SUMMARY:
The purpose of the study is to determine the safety and efficacy of the use of bendamustine in combination with a commonly used combination chemotherapy to treat relapsed and refractory multiple myeloma. The study will be conducted in two phases. Participants in phase I will receive 1 of 4 escalating doses of bendamustine. Once the maximum tolerated dose of bendamustine is determined, phase II of this trial will begin. Participants in phase II will receive the maximum tolerated dose of bendamustine in combination with standard of care chemotherapy.

DETAILED DESCRIPTION:
Multiple myeloma is a multi-organ neoplastic disorder caused by the clonal proliferation of plasma cells. It has an incidence of about 4.5/100,000 per year in the U.S., making it the second most common hematologic malignancy. For many years, alkylating agents have been the backbone of treatment. The combination of melphalan and prednisone was, for many years, the standard of care for patients who were not candidates for autologous transplantation. Melphalan continues to be the primary conditioning agent for autologous transplant,and cyclophosphamide has also gained a foothold in the treatment of this disease.

The introduction of novel agents has fundamentally changed the landscape of treating this disease, although the true effects on survival are not yet known. Immunomodulatory agents and proteosome inhibitors, including thalidomide, lenalidomide and bortezomib have been used in both newly diagnosed and relapsed patients. Currently, there is intense clinical research on the optimal way to combine these novel agents with the traditional backbones of treatment - including alkylators, with one another and, eventually, with the subsequent iterations of these classes of drugs. However, despite the therapeutic excitement surrounding this disease, most patients will relapse and a cure remains an elusive goal.

ELIGIBILITY:
Inclusion Criteria:

* Adults with relapsed and/or refractory myeloma who have received between 1-4 prior lines of therapy
* Must have adequate liver and renal function
* Zubrod Performance Status (ZPS) of 2 or better
* Must have measurable disease

Exclusion Criteria:

* Peripheral neuropathy of grade II or higher
* Thrombocytopenia (platelets less than 50,000/uL)
* Neutropenia (ANC<1000/uL)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.4 X ULN
* Total bilirubin >1.5 X upper limit of normal (ULN)
* Creatinine clearance of less than 45 milliliters per minute (mL/min)
* Patients with HIV
* Patients with active hepatitis
* Pregnant or lactating women
* Individuals of child-bearing potential not using adequate contraception
* Individuals unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-05-05 (Actual); Primary Completion 2014-06-18 (Actual); Study Completion 2014-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Smith, MD, PhD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634
- [Background] Fenk R, Michael M, Zohren F, Graef T, Czibere A, Bruns I, Neumann F, Fenk B, Haas R, Kobbe G. Escalation therapy with bortezomib, dexamethasone and bendamustine for patients with relapsed or refractory multiple myeloma. Leuk Lymphoma. 2007 Dec;48(12):2345-51. doi: 10.1080/10428190701694194. PMID 18067009
- [Background] Harousseau JL, Moreau P. Autologous hematopoietic stem-cell transplantation for multiple myeloma. N Engl J Med. 2009 Jun 18;360(25):2645-54. doi: 10.1056/NEJMct0805626. No abstract available. PMID 19535803
- [Background] Knop S, Straka C, Haen M, Schwedes R, Hebart H, Einsele H. The efficacy and toxicity of bendamustine in recurrent multiple myeloma after high-dose chemotherapy. Haematologica. 2005 Sep;90(9):1287-8. PMID 16154860
- [Background] Kyle RA, Rajkumar SV. Multiple myeloma. Blood. 2008 Mar 15;111(6):2962-72. doi: 10.1182/blood-2007-10-078022. PMID 18332230
- [Background] Lee CK, Barlogie B, Munshi N, Zangari M, Fassas A, Jacobson J, van Rhee F, Cottler-Fox M, Muwalla F, Tricot G. DTPACE: an effective, novel combination chemotherapy with thalidomide for previously treated patients with myeloma. J Clin Oncol. 2003 Jul 15;21(14):2732-9. doi: 10.1200/JCO.2003.01.055. PMID 12860952
- [Background] Palumbo A, Facon T, Sonneveld P, Blade J, Offidani M, Gay F, Moreau P, Waage A, Spencer A, Ludwig H, Boccadoro M, Harousseau JL. Thalidomide for treatment of multiple myeloma: 10 years later. Blood. 2008 Apr 15;111(8):3968-77. doi: 10.1182/blood-2007-10-117457. Epub 2008 Feb 1. PMID 18245666
- [Background] Ponisch W, Mitrou PS, Merkle K, Herold M, Assmann M, Wilhelm G, Dachselt K, Richter P, Schirmer V, Schulze A, Subert R, Harksel B, Grobe N, Stelzer E, Schulze M, Bittrich A, Freund M, Pasold R, Friedrich T, Helbig W, Niederwieser D; East German Study Group of Hematology and Oncology (OSHO). Treatment of bendamustine and prednisone in patients with newly diagnosed multiple myeloma results in superior complete response rate, prolonged time to treatment failure and improved quality of life compared to treatment with melphalan and prednisone--a randomized phase III study of the East German Study Group of Hematology and Oncology (OSHO). J Cancer Res Clin Oncol. 2006 Apr;132(4):205-12. doi: 10.1007/s00432-005-0074-4. Epub 2006 Jan 10. PMID 16402269
- [Background] Ponisch W, Rozanski M, Goldschmidt H, Hoffmann FA, Boldt T, Schwarzer A, Ritter U, Rohrberg R, Schwalbe E, Uhlig J, Zehrfeld T, Schirmer V, Haas A, Kreibich U, Niederwieser D; East German Study Group of Haematology and Oncology (OSHO). Combined bendamustine, prednisolone and thalidomide for refractory or relapsed multiple myeloma after autologous stem-cell transplantation or conventional chemotherapy: results of a Phase I clinical trial. Br J Haematol. 2008 Oct;143(2):191-200. doi: 10.1111/j.1365-2141.2008.07076.x. Epub 2008 Aug 24. PMID 18752593
- [Background] Rajkumar SV, Hayman SR, Lacy MQ, Dispenzieri A, Geyer SM, Kabat B, Zeldenrust SR, Kumar S, Greipp PR, Fonseca R, Lust JA, Russell SJ, Kyle RA, Witzig TE, Gertz MA. Combination therapy with lenalidomide plus dexamethasone (Rev/Dex) for newly diagnosed myeloma. Blood. 2005 Dec 15;106(13):4050-3. doi: 10.1182/blood-2005-07-2817. Epub 2005 Aug 23. PMID 16118317
- [Background] Richardson PG, Sonneveld P, Schuster MW, Irwin D, Stadtmauer EA, Facon T, Harousseau JL, Ben-Yehuda D, Lonial S, Goldschmidt H, Reece D, San-Miguel JF, Blade J, Boccadoro M, Cavenagh J, Dalton WS, Boral AL, Esseltine DL, Porter JB, Schenkein D, Anderson KC; Assessment of Proteasome Inhibition for Extending Remissions (APEX) Investigators. Bortezomib or high-dose dexamethasone for relapsed multiple myeloma. N Engl J Med. 2005 Jun 16;352(24):2487-98. doi: 10.1056/NEJMoa043445. PMID 15958804
- [Background] San-Miguel J, Harousseau JL, Joshua D, Anderson KC. Individualizing treatment of patients with myeloma in the era of novel agents. J Clin Oncol. 2008 Jun 1;26(16):2761-6. doi: 10.1200/JCO.2007.15.2546. Epub 2008 Apr 21. PMID 18427148
- [Background] San Miguel JF, Schlag R, Khuageva NK, Dimopoulos MA, Shpilberg O, Kropff M, Spicka I, Petrucci MT, Palumbo A, Samoilova OS, Dmoszynska A, Abdulkadyrov KM, Schots R, Jiang B, Mateos MV, Anderson KC, Esseltine DL, Liu K, Cakana A, van de Velde H, Richardson PG; VISTA Trial Investigators. Bortezomib plus melphalan and prednisone for initial treatment of multiple myeloma. N Engl J Med. 2008 Aug 28;359(9):906-17. doi: 10.1056/NEJMoa0801479. PMID 18753647
- [Background] Adams J, Palombella VJ, Sausville EA, Johnson J, Destree A, Lazarus DD, Maas J, Pien CS, Prakash S, Elliott PJ. Proteasome inhibitors: a novel class of potent and effective antitumor agents. Cancer Res. 1999 Jun 1;59(11):2615-22. PMID 10363983
- [Background] Teicher BA, Ara G, Herbst R, Palombella VJ, Adams J. The proteasome inhibitor PS-341 in cancer therapy. Clin Cancer Res. 1999 Sep;5(9):2638-45. PMID 10499643
- [Background] Cusack JC Jr, Liu R, Houston M, Abendroth K, Elliott PJ, Adams J, Baldwin AS Jr. Enhanced chemosensitivity to CPT-11 with proteasome inhibitor PS-341: implications for systemic nuclear factor-kappaB inhibition. Cancer Res. 2001 May 1;61(9):3535-40. PMID 11325813
- [Background] LeBlanc R, Catley LP, Hideshima T, Lentzsch S, Mitsiades CS, Mitsiades N, Neuberg D, Goloubeva O, Pien CS, Adams J, Gupta D, Richardson PG, Munshi NC, Anderson KC. Proteasome inhibitor PS-341 inhibits human myeloma cell growth in vivo and prolongs survival in a murine model. Cancer Res. 2002 Sep 1;62(17):4996-5000. PMID 12208752
- [Background] Williams S, Pettaway C, Song R, Papandreou C, Logothetis C, McConkey DJ. Differential effects of the proteasome inhibitor bortezomib on apoptosis and angiogenesis in human prostate tumor xenografts. Mol Cancer Ther. 2003 Sep;2(9):835-43. PMID 14555702
- [Background] Nawrocki ST, Bruns CJ, Harbison MT, Bold RJ, Gotsch BS, Abbruzzese JL, Elliott P, Adams J, McConkey DJ. Effects of the proteasome inhibitor PS-341 on apoptosis and angiogenesis in orthotopic human pancreatic tumor xenografts. Mol Cancer Ther. 2002 Dec;1(14):1243-53. PMID 12516957
- [Background] Satou Y, Nosaka K, Koya Y, Yasunaga JI, Toyokuni S, Matsuoka M. Proteasome inhibitor, bortezomib, potently inhibits the growth of adult T-cell leukemia cells both in vivo and in vitro. Leukemia. 2004 Aug;18(8):1357-63. doi: 10.1038/sj.leu.2403400. PMID 15190257
- [Background] Boccadoro M, Morgan G, Cavenagh J. Preclinical evaluation of the proteasome inhibitor bortezomib in cancer therapy. Cancer Cell Int. 2005 Jun 1;5(1):18. doi: 10.1186/1475-2867-5-18. PMID 15929791
- [Background] Goel A, Dispenzieri A, Geyer SM, Greiner S, Peng KW, Russell SJ. Synergistic activity of the proteasome inhibitor PS-341 with non-myeloablative 153-Sm-EDTMP skeletally targeted radiotherapy in an orthotopic model of multiple myeloma. Blood. 2006 May 15;107(10):4063-70. doi: 10.1182/blood-2005-09-3870. Epub 2006 Jan 19. PMID 16424391
- [Background] Mitsiades N, Mitsiades CS, Richardson PG, Poulaki V, Tai YT, Chauhan D, Fanourakis G, Gu X, Bailey C, Joseph M, Libermann TA, Schlossman R, Munshi NC, Hideshima T, Anderson KC. The proteasome inhibitor PS-341 potentiates sensitivity of multiple myeloma cells to conventional chemotherapeutic agents: therapeutic applications. Blood. 2003 Mar 15;101(6):2377-80. doi: 10.1182/blood-2002-06-1768. Epub 2002 Nov 7. PMID 12424198
- [Background] Sayers TJ, Brooks AD, Koh CY, Ma W, Seki N, Raziuddin A, Blazar BR, Zhang X, Elliott PJ, Murphy WJ. The proteasome inhibitor PS-341 sensitizes neoplastic cells to TRAIL-mediated apoptosis by reducing levels of c-FLIP. Blood. 2003 Jul 1;102(1):303-10. doi: 10.1182/blood-2002-09-2975. Epub 2003 Mar 13. PMID 12637321
- [Background] Yu C, Rahmani M, Conrad D, Subler M, Dent P, Grant S. The proteasome inhibitor bortezomib interacts synergistically with histone deacetylase inhibitors to induce apoptosis in Bcr/Abl+ cells sensitive and resistant to STI571. Blood. 2003 Nov 15;102(10):3765-74. doi: 10.1182/blood-2003-03-0737. Epub 2003 Jul 31. PMID 12893773
- [Background] O'Connor OA, Smith EA, Toner LE, Teruya-Feldstein J, Frankel S, Rolfe M, Wei X, Liu S, Marcucci G, Chan KK, Chanan-Khan A. The combination of the proteasome inhibitor bortezomib and the bcl-2 antisense molecule oblimersen sensitizes human B-cell lymphomas to cyclophosphamide. Clin Cancer Res. 2006 May 1;12(9):2902-11. doi: 10.1158/1078-0432.CCR-05-0308. PMID 16675587
- [Background] David E, Sun SY, Waller EK, Chen J, Khuri FR, Lonial S. The combination of the farnesyl transferase inhibitor lonafarnib and the proteasome inhibitor bortezomib induces synergistic apoptosis in human myeloma cells that is associated with down-regulation of p-AKT. Blood. 2005 Dec 15;106(13):4322-9. doi: 10.1182/blood-2005-06-2584. Epub 2005 Aug 23. PMID 16118318
- [Background] Hideshima T, Richardson P, Chauhan D, Palombella VJ, Elliott PJ, Adams J, Anderson KC. The proteasome inhibitor PS-341 inhibits growth, induces apoptosis, and overcomes drug resistance in human multiple myeloma cells. Cancer Res. 2001 Apr 1;61(7):3071-6. PMID 11306489
- [Background] Obeng EA, Carlson LM, Gutman DM, Harrington WJ Jr, Lee KP, Boise LH. Proteasome inhibitors induce a terminal unfolded protein response in multiple myeloma cells. Blood. 2006 Jun 15;107(12):4907-16. doi: 10.1182/blood-2005-08-3531. Epub 2006 Feb 28. PMID 16507771
- [Background] Ling YH, Liebes L, Ng B, Buckley M, Elliott PJ, Adams J, Jiang JD, Muggia FM, Perez-Soler R. PS-341, a novel proteasome inhibitor, induces Bcl-2 phosphorylation and cleavage in association with G2-M phase arrest and apoptosis. Mol Cancer Ther. 2002 Aug;1(10):841-9. PMID 12492117
- [Background] Yang Y, Ikezoe T, Saito T, Kobayashi M, Koeffler HP, Taguchi H. Proteasome inhibitor PS-341 induces growth arrest and apoptosis of non-small cell lung cancer cells via the JNK/c-Jun/AP-1 signaling. Cancer Sci. 2004 Feb;95(2):176-80. doi: 10.1111/j.1349-7006.2004.tb03200.x. PMID 14965369
- [Background] Kaluz S, Kaluzova M, Stanbridge EJ. Proteasomal inhibition attenuates transcriptional activity of hypoxia-inducible factor 1 (HIF-1) via specific effect on the HIF-1alpha C-terminal activation domain. Mol Cell Biol. 2006 Aug;26(15):5895-907. doi: 10.1128/MCB.00552-06. PMID 16847340
- [Background] An WG, Hwang SG, Trepel JB, Blagosklonny MV. Protease inhibitor-induced apoptosis: accumulation of wt p53, p21WAF1/CIP1, and induction of apoptosis are independent markers of proteasome inhibition. Leukemia. 2000 Jul;14(7):1276-83. doi: 10.1038/sj.leu.2401812. PMID 10914553
- [Background] Roccaro AM, Hideshima T, Raje N, Kumar S, Ishitsuka K, Yasui H, Shiraishi N, Ribatti D, Nico B, Vacca A, Dammacco F, Richardson PG, Anderson KC. Bortezomib mediates antiangiogenesis in multiple myeloma via direct and indirect effects on endothelial cells. Cancer Res. 2006 Jan 1;66(1):184-91. doi: 10.1158/0008-5472.CAN-05-1195. PMID 16397231
- [Background] Mitsiades N, Mitsiades CS, Poulaki V, Chauhan D, Fanourakis G, Gu X, Bailey C, Joseph M, Libermann TA, Treon SP, Munshi NC, Richardson PG, Hideshima T, Anderson KC. Molecular sequelae of proteasome inhibition in human multiple myeloma cells. Proc Natl Acad Sci U S A. 2002 Oct 29;99(22):14374-9. doi: 10.1073/pnas.202445099. Epub 2002 Oct 21. PMID 12391322
- [Background] Orlowski RZ, Stinchcombe TE, Mitchell BS, Shea TC, Baldwin AS, Stahl S, Adams J, Esseltine DL, Elliott PJ, Pien CS, Guerciolini R, Anderson JK, Depcik-Smith ND, Bhagat R, Lehman MJ, Novick SC, O'Connor OA, Soignet SL. Phase I trial of the proteasome inhibitor PS-341 in patients with refractory hematologic malignancies. J Clin Oncol. 2002 Nov 15;20(22):4420-7. doi: 10.1200/JCO.2002.01.133. PMID 12431963
- [Background] Aghajanian C, Soignet S, Dizon DS, Pien CS, Adams J, Elliott PJ, Sabbatini P, Miller V, Hensley ML, Pezzulli S, Canales C, Daud A, Spriggs DR. A phase I trial of the novel proteasome inhibitor PS341 in advanced solid tumor malignancies. Clin Cancer Res. 2002 Aug;8(8):2505-11. PMID 12171876
- [Background] Papandreou CN, Daliani DD, Nix D, Yang H, Madden T, Wang X, Pien CS, Millikan RE, Tu SM, Pagliaro L, Kim J, Adams J, Elliott P, Esseltine D, Petrusich A, Dieringer P, Perez C, Logothetis CJ. Phase I trial of the proteasome inhibitor bortezomib in patients with advanced solid tumors with observations in androgen-independent prostate cancer. J Clin Oncol. 2004 Jun 1;22(11):2108-21. doi: 10.1200/JCO.2004.02.106. PMID 15169797
- [Background] Dimopoulos MA, Anagnostopoulos A, Kyrtsonis MC, Castritis E, Bitsaktsis A, Pangalis GA. Treatment of relapsed or refractory Waldenstrom's macroglobulinemia with bortezomib. Haematologica. 2005 Dec;90(12):1655-8. PMID 16330439
- [Background] Jagannath S, Barlogie B, Berenson J, Siegel D, Irwin D, Richardson PG, Niesvizky R, Alexanian R, Limentani SA, Alsina M, Adams J, Kauffman M, Esseltine DL, Schenkein DP, Anderson KC. A phase 2 study of two doses of bortezomib in relapsed or refractory myeloma. Br J Haematol. 2004 Oct;127(2):165-72. doi: 10.1111/j.1365-2141.2004.05188.x. PMID 15461622
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- [Background] Fisher RI, Bernstein SH, Kahl BS, Djulbegovic B, Robertson MJ, de Vos S, Epner E, Krishnan A, Leonard JP, Lonial S, Stadtmauer EA, O'Connor OA, Shi H, Boral AL, Goy A. Multicenter phase II study of bortezomib in patients with relapsed or refractory mantle cell lymphoma. J Clin Oncol. 2006 Oct 20;24(30):4867-74. doi: 10.1200/JCO.2006.07.9665. Epub 2006 Sep 25. PMID 17001068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from May 2011 through April 2014 (36 months) from the Cardinal Bernardin Cancer Center at Loyola University Medical Center
Pre-assignment Details: There are no pre-assignment details to report
Period: Overall Study
Arm/Group | Bendamustine
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all participants who signed an informed consent document
Arm/Group | Bendamustine
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing a Toxicity
Description: The number of patients experiencing at least one toxicity at the lowest dose of bendamustine. A toxicity is defined as one or more of the following: Upper respiratory infection; anemia; thrombocytopenia; neutropenia; shortness of breath on exertion; decreased appetite; nausea; neuropathy; anxiety; arthritis; and hypercalcemia.
Time Frame: 21 days
Population: No patients were analyzed as study was terminated early after external sponsor withdrew support. Therefore, data necessary for planned analyses were not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine
Number analyzed (Participants) | 3
Participants
  Experienced no toxicities | 0
  Experienced at least one toxicity | 3

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from November 2011 through June 2014 (32 months)
Arm/Group | Bendamustine
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=3)
Upper respiratory infection (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Shortness of Breath on Exertion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decreased appetite (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Arthritis (Endocrine disorders) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial terminated in June 2014 when Celgene could no longer supply lenalidomide for the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes